CLINICAL TRIAL: NCT01783392
Title: Peripheral Electrical Stimulation for the Treatment of Overactive Bladder
Acronym: PESTOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH16245
Record Dates: First submitted 2013-01-23; First posted 2013-02-04 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Idiopathic Overactive Bladder
Keywords: overactive bladder; transcutaneous posterior tibial nerve stimulation; placebo PTNS
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Transcutaneous Electric Nerve Stimulation

ARMS (3):
- Unilateral Posterior Tibial Nerve Stimulation (Active Comparator): Transcutaneous posterior tibial nerve stimulation applied 40 minutes every day for a duration of 4 weeks. The patient places the cathode electrode above, and the anode electrode behind, the medial malleolus, over the posterior tibial nerve and sets the stimulation intensity to a comfortable level.
  Interventions: Procedure: Transcutaneous Electrical Nerve Stimulation
- Bilateral Posterior Tibial Nerve Stimulation (Active Comparator): Transcutaneous posterior tibial nerve stimulation applied 40 minutes every day for a duration of 4 weeks. The patient places the cathode electrode above, and the anode electrode behind, the medial malleolus, over the posterior tibial nerve on both legs and sets the stimulation intensity to a comfortable level.
  Interventions: Procedure: Transcutaneous Electrical Nerve Stimulation
- Shoulder stimulation (Active Comparator): Stimulation applied 40 minutes every day for a duration of 4 weeks. The patient places the cathode and the anode electrodes on the lateral side of the left shoulder.
  Interventions: Procedure: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Procedure: Transcutaneous Electrical Nerve Stimulation

SUMMARY:
This clinical trial testing three different sites of transcutaneous electrical nerve stimulation for the treatment of overactive bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, at least 18 years of age
* Documented symptoms of idiopathic overactive bladder for at least 3 months
* Failure on primary OAB treatment, such as behavior modification or fluid/diet management
* Patients can remain on stable medication
* Willing and capable of understanding and complying with all requirements of the protocol
* Signed Informed Consent to participate in the study after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* Urinary retention or post voiding residual greater than 100 ml
* Clinically significant bladder outlet obstruction
* Stress predominant mixed urinary incontinence
* Neurological disease affecting urinary bladder function, including but not limited to Parkinson's disease, multiple sclerosis, stroke, spinal cord injury.
* Pelvic surgery (such as sub-urethral sling, pelvic floor repair) within the past 6 months
* Denovo OAB following pelvic surgery sub-urethral sling Intravesical or urethral sphincter Botulinum Toxin Type A injections within the past 6 months
* Percutaneous Tibial Nerve Stimulation (PTNS) therapy for overactive bladder within the past 6 months
* Any form of electric stimulation to the pelvis or lower limbs within 4 weeks
* Vaginal prolapse greater than Stage II in the anterior compartment of the vagina using International Continence Society (ICS) Pelvic Organ ProlapseQuantification (POPQ) criteria.
* Prior periurethral or transurethral bulking agent injections for bladder problems within the past 12 months.
* History of pelvic radiation therapy
* Any skin conditions affecting treatment sites
* Lacking dexterity to properly utilize the components of the stimulator system.
* Presence of an implanted electro-medical device (e.g. pacemaker, defibrillator, InterStim®, etc.),
* Pregnant, nursing, suspected to be pregnant (by urine pregnancy method), or plans to become pregnant during the course of the study.
* Recurrent Urinary Tract Infections UTI (>3 UTI's in the past year)
* History of, or current, lower tract genitourinary malignancies
* Any clinically significant systemic disease or condition that in the opinion of the Investigator would make the patient unsuitable for the study
* Any other clinical trial within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in frequency of voiding | baseline, 4 weeks
  The change of urinary frequency from baseline to after 4 weeks of the treatment, measured by a 3 days bladder diary.
Change in Patient Perception of Bladder Condition (PPBC) | baseline, 4 weeks
  Change in the patient's bladder condition based on the PPBC questionaire from baseline to after 4 weeks of the treatment.

SECONDARY OUTCOMES:
Changes in symptom severity score and health-related quality of life score (HRQL) based on OAB-questionnaire | baseline, 4 weeks
  Change in symptom severity score and HRQL score from baseline to after 4weeks of the treatment.
Changes in the mental/physical scores of RAND36 | baseline, 4 weeks
Change in urinary symptoms score and bother symptom score based on the ICIQ-OAB questionnaire | baseline, 4 weeks
  Change in urinary symptoms score and bother symptom score based on the ICIQ-OAB questionnaire from baseline to after 4 weeks of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chapple, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS foundation Trust, Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom